CLINICAL TRIAL: NCT05714670
Title: The Effect of Curcumin on the Clinical Outcome of Pediatric Patients with Active Lupus Nephritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, sujoud hosam, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHDIRB2020110301REC121
Record Dates: First submitted 2023-01-19; First posted 2023-02-06 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-01

CONDITIONS: Lupus Nephritis; SLE Nephritis
Keywords: curcumin; herbal medicine; lupus nephritis; paediatric onset SLE
MeSH Terms: conditions — Lupus Nephritis | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: Group I: patients will receive the studied drug orally in addition to their standard treatment for three months.
  Group II: patients will receive only their standard treatment for three months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- standard of care (No Intervention): patients will receive oral MMF initial dose of 1200 mg/m2/day, no more than 2000 mg/day, increased to 1800 mg/m2/day, no more than 3000 mg/day, if response is not good + corticosteroid protocols are: intravenous pulse of methylprednisolone (30 mg/kg/dose for three consecutive days, no more than de 1000 mg/dose), followed by oral prednisolone/prednisone (0.5-1.0 mg/kg/day); or high dosage oral prednisone/prednisolone (1-2 mg/kg/day, no more than 60 mg/day) + hydroxychloroquine 4.0-5.5 mg/kg/day second regimen: low-dose intravenous cyclophosphamide (CY) (total dose 3 g over 3 months) -monthly pulses 0.5-1 g/m2- in combination with glucocorticoids
- Curcumin Oral Capsule group (Experimental): patients will receive oral 1000 mg of curcumin capsules daily in addition to their standard treatment for three months.
  Standard treatment includes: oral MMF initial dose of 1200 mg/m2/day, no more than 2000 m g/day, increased to 1800 mg/m2/day, no more than 3000 mg/day, if response is not good + corticosteroid protocols are: intravenous pulse of methylprednisolone (30 mg/kg/dose for three consecutive days, no more than de 1000 mg/dose), followed by oral prednisolone/prednisone (0.5-1.0 mg/kg/day); or high dosage oral prednisone/prednisolone (1-2 mg/kg/day, no more than 60 mg/day) + hydroxychloroquine 4.0-5.5 mg/kg/day
  second regimen: low-dose intravenous cyclophosphamide (CY) (total dose 3 g over 3 months) -monthly pulses 0.5-1 g/m2- in combination with glucocorticoids
  Interventions: Drug: Curcumin Oral Capsule

INTERVENTIONS:
Drug: Curcumin Oral Capsule — Curcumin 1000 mg Oral Capsule beside the standard of care
  Other Names: Turmeric
  Arms: Curcumin Oral Capsule group

SUMMARY:
Pediatric Lupus nephritis which is a sever and common complication to childhood onset systemic lupus erythematous is an aggressive inflammatory process triggered by the deposition of antigen-antibody complex in kidney tissue. The complex stimulates production of multiple immune cells, activating Inflammasome NLRP3 that plays massive role in stimulating various cytokines like IL-6. The inflammation also causes elevation in proteinuria and serum creatinine levels beside other inflammatory markers elevation (CRP )and (ESR). These children are treated with a standard regimen consists of an immunomodulator (mycophenolate mofetil) with strong steroid anti-inflammatory and also hydroxychloroquine is added to the regimen to decrease the intensity of the flares and management of arthritis symptoms. In our study we are introducing a powerful antioxidant and anti-inflammatory drug with nephroprotective benefits which is curcumin capsules. The drug showed success in managing different autoimmune and inflammatory diseases as rheumatoid arthritis and Crohn's disease, it also showed dramatic improvement in lupus nephritis models in previous experimental study. The study primary outcome is will be the composite of the effect of curcumin on Urine protein-to-creatinine ratio and NLPR3 Inflammasome levels in blood. Patients meeting the study inclusion criteria will be educated firmly about the disease details and all information about the drug, then will be randomly assigned to one of two groups, the first group receiving the standard therapy only while the second one receiving the standard therapy beside the curcumin 1000 mg capsules orally daily, a third small group of healthy children as a control for normal inflammasome levels. Patients in the first two groups will undergo baseline evaluation at the beginning of the study including Patients' demographic data, anthropometric measures and medication history. Moreover, collecting patients' medical history which includes Duration of systemic lupus, Duration of lupus nephritis, other organs involvement, past and current medical condition or prescribed and OTC medications. Laboratory Evaluation and renal function assessment will include Inflammasome levels in blood using ELISA technique using Human NLRP3 ELISA Kit, Serum creatinine levels, Protein in urine levels, estimated glomerular filtration rate (eGFR) using Original Schwartz Equations, Inflammatory biomarkers (ESR, CRP), anti-ds DNA, anti-ANA DNA and evaluating Hematuria. Baseline Clinical evaluation includes Blood pressure measurement and Kidney structural damage evaluation via biopsy. Then patients will be followed up monthly for three months for assessing Patient Compliance with the prescribed medication regimens and the study drug, Occurrence of side effect graded using monitoring of side effects scale (MOSES) and checking for Allergic reactions against the drug. After the three months, all patients will be reassessed for all laboratory and clinical evaluations. finally results will be statistically analyzed Statistical analysis will be done using SPSS statistical software package

ELIGIBILITY:
Inclusion Criteria:

* 1- Lupus nephritis patients both genders aged 16 or younger 2- Biopsy specimens confirmed active lesions or active and chronic lesions defined as nephritis according to WHO classification 3- Children on standard treatment (mycophenolate mofetil + hydroxychloroquine + steroids) 4- Children on another standard regimen: low-dose intravenous cyclophosphamide (CY) (total dose 3 g over 3 months) -monthly pulses 0.5-1 g/m2- in combination with glucocorticoids

Exclusion Criteria:

1. Dialysis or B cell-targeted therapy (including belimumab) within the preceding year
2. Patients with other comorbidities
3. Smokers
4. Previous failures of both MMF and CYC induction therapy,
5. Estimated glomerular filtration rate (eGFR) of less than 30 ml/min per 1.73 m2 of body surface area.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
chang is being assessed in Urine protein-to-creatinine ratio from baseline | baseline and week12
  urine sample will be examined for albumin levels and creatinine levels, normal ratio for paediatrics is less than 0.25
change is being assessed in NLPR3 Inflammasome serum levels from baseline | baseline and week12
  serum sample will be examined for NLRP3 inflammasome levels and how it is affected by the tested drug

SECONDARY OUTCOMES:
Erythrocyte sedimentation rate | baseline, week 4, week 8 and week 12
  blood sample is examined for ESR level
C-reactive protein | baseline, week 4, week 8 and week 12
  blood sample is examined for CRP level
Anti-ANA DNA | baseline and week 12
  antinuclear antibody

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatients Clinic of Pediatric Rheumatology department - Children's Hospital, Ain Shams University, Cairo, Egypt., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No